CLINICAL TRIAL: NCT04064879
Title: The Use of Autologous Mesenchymal Stem Cell Preparation for Treatment of Refractory Migraine
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Pending FDA approval
Sponsor: Neurological Associates of West Los Angeles (Other)
Collaborators: Cell Surgical Network Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICSS-2018-014
Record Dates: First submitted 2019-08-19; First posted 2019-08-22 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Chronic Migraine, Headache
MeSH Terms: conditions — Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deployment of AD-SVF (Experimental): Administration of autologous adipose derived SVF
  Interventions: Other: AD-SVF

INTERVENTIONS:
Other: AD-SVF — Intravenous, intra-articular, and soft tissue injection delivery of SVF. Target regions include forehead, temporal, and suboccipital regions.
  Other Names: Mesenchymal Stem Cells

SUMMARY:
The present study is being undertaken as a phase I study to determine the safety and feasibility of using adipose derived mesenchymal stem cell preparations (MSC) for treatment of CM. Intravenous and locally targeted stem cell treatment have already been reported in the context of treating various chronic pain conditions with early evidence of efficacy and a good safety profile. The treatment of CM is based on the model for treatment with botulinum where superficial facial and cranial injections are utilized. In addition, stem cells can be given intravenously as well.

DETAILED DESCRIPTION:
Chronic migraine (CM) is a disabling complex neurological disorder recognized as a complication of migraine in the the International Classification of Headache Disorders. Patients with CM experience headache on 15 days per month. CM is associated with significant disability and reduced health-related quality of life. Approximately 1.3% to 2.4% of the general population suffers from CM, and one in five CM sufferers cannot work because this condition impacts their ability to lead productive lives. CM is frequently complicated by overuse of acute pain medications. Some drugs have regulatory approval for migraine prophylaxis; none are approved specifically for CM prophylaxis although recently, botulinum injection has been FDA approved for CM treatment with marginal treatment effects with many patients failing to have complete remission. The present study is being undertaken as a phase I study to determine the safety and feasibility of using adipose derived mesenchymal stem cell preparations (MSC) for treatment of CM.

ELIGIBILITY:
Inclusion Criteria:

* Patients must exhibit symptoms that satisfy criteria of Chronic Migraine (e.g., experiencing headaches at least 15 days per month to a degree that is associated with significant disability and reduced health-related quality of life).

Exclusion Criteria:

* Advanced stages of any terminal illness or active cancer that requires chemotherapy.
* Pregnancy, women who may become pregnant or are breastfeeding.
* Bleeding disorder, untreated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2023-08-15 (Estimated); Study Completion 2023-08-16 (Estimated)

PRIMARY OUTCOMES:
Adverse Event Reporting | Throughout study duration (Baseline through 36 months)
  Any participants with adverse events suspected to be related to either SVF deployment or the lipo-harvesting procedure were noted and reported immediately.

SECONDARY OUTCOMES:
Headache Diary | 2 months
  Headache pain is scored on a range from 0 'no pain' to 10 'worst pain ever.' Patients reported the number of headaches total per month (each diary has a total possible number of 31 entries).Total score is calculated by adding the sum score of each headache (maximum possible = 310). Clinical improvement was noted for patients whose scores improved by at least 20%.
Headache Impact Test (HIT-6) | 2 months
  The HIT-6 is a self-report questionnaire consisting of 6 questions, with qualitative answers ranging from "never," "rarely," "sometimes," "very often," and "always" to describe the frequency and impact of headaches on patient lives. Answers correspond with point values as following: never = 6 points, rarely = 8 points, sometimes = 10 points, very often = 11 points, & always = 13 points. A total score of 50 or more indicates severe disability related to headaches. Clinical improvement was noted for patients who reported at least a 20% decrease in their scores from baseline.
Headache Diary | 6 months
  Headache pain is scored on a range from 0 'no pain' to 10 'worst pain ever.' Patients reported the number of headaches total per month (each diary has a total possible number of 31 entries).Total score is calculated by adding the sum score of each headache (maximum possible = 310). Clinical improvement was noted for patients whose scores improved by at least 20% from baseline.
Headache Impact Test (HIT-6) | 6 months
  The HIT-6 is a self-report questionnaire consisting of 6 questions, with qualitative answers ranging from "never," "rarely," "sometimes," "very often," and "always" to describe the frequency and impact of headaches on patient lives. Answers correspond with point values as following: never = 6 points, rarely = 8 points, sometimes = 10 points, very often = 11 points, & always = 13 points. A total score of 50 or more indicates severe disability related to headaches. Clinical improvement was noted for patients who reported at least a 20% decrease in their scores from baseline.
Headache Diary | 1 year
  Headache pain is scored on a range from 0 'no pain' to 10 'worst pain ever.' Patients reported the number of headaches total per month (each diary has a total possible number of 31 entries).Total score is calculated by adding the sum score of each headache (maximum possible = 310). Clinical improvement was noted for patients whose scores improved by at least 20% from baseline.
Headache Impact Test (HIT-6) | 1 year
  The HIT-6 is a self-report questionnaire consisting of 6 questions, with qualitative answers ranging from "never," "rarely," "sometimes," "very often," and "always" to describe the frequency and impact of headaches on patient lives. Answers correspond with point values as following: never = 6 points, rarely = 8 points, sometimes = 10 points, very often = 11 points, & always = 13 points. A total score of 50 or more indicates severe disability related to headaches. Clinical improvement was noted for patients who reported at least a 20% decrease in their scores from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon E Jordan, MD, FAAN, Principal Investigator — Neurological Associates of West Los Angeles
Locations (1):
- Neurological Associates of West Los Angeles, Santa Monica, California, United States

REFERENCES:
- [Background] Headache Classification Subcommittee of the International Headache Society. The International Classification of Headache Disorders: 2nd edition. Cephalalgia. 2004;24 Suppl 1:9-160. doi: 10.1111/j.1468-2982.2003.00824.x. No abstract available. PMID 14979299
- [Background] Headache Classification Committee; Olesen J, Bousser MG, Diener HC, Dodick D, First M, Goadsby PJ, Gobel H, Lainez MJ, Lance JW, Lipton RB, Nappi G, Sakai F, Schoenen J, Silberstein SD, Steiner TJ. New appendix criteria open for a broader concept of chronic migraine. Cephalalgia. 2006 Jun;26(6):742-6. doi: 10.1111/j.1468-2982.2006.01172.x. PMID 16686915
- [Background] Dodick DW. Clinical practice. Chronic daily headache. N Engl J Med. 2006 Jan 12;354(2):158-65. doi: 10.1056/NEJMcp042897. No abstract available. PMID 16407511
- [Background] Bigal ME, Serrano D, Reed M, Lipton RB. Chronic migraine in the population: burden, diagnosis, and satisfaction with treatment. Neurology. 2008 Aug 19;71(8):559-66. doi: 10.1212/01.wnl.0000323925.29520.e7. PMID 18711108
- [Background] Castillo J, Munoz P, Guitera V, Pascual J. Kaplan Award 1998. Epidemiology of chronic daily headache in the general population. Headache. 1999 Mar;39(3):190-6. doi: 10.1046/j.1526-4610.1999.3903190.x. PMID 15613213
- [Background] Scher AI, Stewart WF, Liberman J, Lipton RB. Prevalence of frequent headache in a population sample. Headache. 1998 Jul-Aug;38(7):497-506. doi: 10.1046/j.1526-4610.1998.3807497.x. PMID 15613165
- [Background] Lanteri-Minet M, Auray JP, El Hasnaoui A, Dartigues JF, Duru G, Henry P, Lucas C, Pradalier A, Chazot G, Gaudin AF. Prevalence and description of chronic daily headache in the general population in France. Pain. 2003 Mar;102(1-2):143-9. doi: 10.1016/s0304-3959(02)00348-2. PMID 12620605
- [Background] Buse DC, Manack A, Serrano D, Turkel C, Lipton RB. Sociodemographic and comorbidity profiles of chronic migraine and episodic migraine sufferers. J Neurol Neurosurg Psychiatry. 2010 Apr;81(4):428-32. doi: 10.1136/jnnp.2009.192492. Epub 2010 Feb 17. PMID 20164501
- [Background] Diener HC, Limmroth V. Medication-overuse headache: a worldwide problem. Lancet Neurol. 2004 Aug;3(8):475-83. doi: 10.1016/S1474-4422(04)00824-5. PMID 15261608
- [Background] Bigal ME, Lipton RB, Tepper SJ, Rapoport AM, Sheftell FD. Primary chronic daily headache and its subtypes in adolescents and adults. Neurology. 2004 Sep 14;63(5):843-7. doi: 10.1212/01.wnl.0000137039.08724.18. PMID 15365134
- [Background] Lipton RB, Bigal ME. Chronic daily headache: is analgesic overuse a cause or a consequence? Neurology. 2003 Jul 22;61(2):154-5. doi: 10.1212/wnl.61.2.154. No abstract available. PMID 12874389
- [Background] Dodick DW, Turkel CC, Degryse RE, Aurora SK, Silberstein SD, Lipton RB, Diener HC, Brin MF. OnabotulinumtoxinA for treatment of chronic migraine: a response. Headache. 2011 Jun;51(6):1005-8. doi: 10.1111/j.1526-4610.2011.01925.x. Epub 2011 May 17. No abstract available. PMID 21592099